CLINICAL TRIAL: NCT03645525
Title: Intratracheal Umbilical Cord-derived Mesenchymal Stem Cell for the Treatment of Bronchopulmonary Dysplasia (BPD)
Acronym: IUMTB
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The certification of cell-based treatment in the settings need to be updated.
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EKYYIUMTB
Record Dates: First submitted 2018-08-16; First posted 2018-08-24 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary Dysplasia; Mesenchymal stem cell
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal stem cell (Experimental): Human Umbilical Cord-derived Mesenchymal stem cell in the saline
  Interventions: Drug: Human Umbilical Cord-derived Mesenchymal stem cell
- placebo (Placebo Comparator): saline without mesenchymal stem cell
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Human Umbilical Cord-derived Mesenchymal stem cell — The Human Umbilical Cord-derived Mesenchymal stem cells suspension (2×10^7/kg per KG of the infant 's weight ) will be instilled once through a catheter into the infant' s endotracheal tube
  Arms: Mesenchymal stem cell
Drug: placebo — saline
  Arms: placebo

SUMMARY:
Umbilical Cord-derived Mesenchymal stem cell has been proven effective in the experimental bronchopulmonary dysplasia (BPD).A multi-center study was designed to evaluate the safety and efficacy of the cellular therapy in extremely preterm infants at high risk for BPD.

DETAILED DESCRIPTION:
Brochopulmonary dysplasia is a severe chronic lung disease in extremely preterm infants. The morbidity of BPD is increasing in CHINA. The preventive and therapy methods of BPD are still lacking.

Umbilical Cord-derived Mesenchymal stem cell has been proven effective in the experimental bronchopulmonary dysplasia (BPD). A multi-center study was designed to evaluate the safety and efficacy of the cellular therapy in extremely preterm infants at high risk for BPD.

ELIGIBILITY:
Inclusion Criteria:

* Extremely preterm infants who remain on mechanic ventilator after 2 weeks of postnatal age
* Extremely preterm infants with a X-ray sign of BPD after 2 weeks of postnatal age

Exclusion Criteria:

* Patients with severe congenital diseases
* Patients with IVH more than 3 grade
* Patients with severe sepsis
* Patients with active pulmonary hemorrhage

Ages: 2 Weeks to 3 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Oxygen requirement 3 days after transplantation | 3 days
  Temporal profiles of the fraction of inspiration oxygen 3 days after transplantation, the tolerable required oxygen ，which is the minimum fraction of inspiration oxygen in which the participants has a stable SpO2 (90%-95%), measured in %

SECONDARY OUTCOMES:
Oxygen requirement 7 days after transplantation | 7 days
  Temporal profiles of the fraction of inspiration oxygen 7 days after transplantation, the tolerable required oxygen ，which is the minimum fraction of inspiration oxygen in which the participants has a stable SpO2 (90%-95%), measured in %
Duration of ventilator dependence | up to 36 weeks PMA
  The duration from transplantation to weaning from ventilator
Incidence of severe BPD | up to 36 weeks PMA
  percentage of participants with severe BPD ,diagnosed at 36 weeks PMA
Survival rate | up to 36 weeks PMA
  Percentage of participants who survived up to 36 weeks PMA
Temperature | 3 days
  Temporal profiles of temperature
Heart rate | 3 days
  Temporal profiles of heart rate
Respiratory rate | 3 days
  Temporal profiles of respiratory rate
Duration of CPAP treatment | up to 36 weeks PMA
  Duration of CPAP treatment
Percentage of participants treated with steroids for weaning from ventilator | up to 36 weeks PMA
  Percentage of participants treated with steroids for weaning from ventilator
Growth velocity (Z-score) | up to 36 weeks PMA
  percentile for body weight, height, and head circumference
bronohoalveolar lavage (BAL) cytokine level | 7 days
  BAL were collected 7 days after transplantation for cytokine (IL-6，IL-8，TNF-α，TGF-β,VEGF,HGF) level examination, measured in pg/ml
The severity of BPD in X-ray patterns | 7 days
  A chest X-ray was performed in participants before and after transplantation. The severity of BPD (mild，moderate，severe) was assessed by a single radiographic doctor who is blind about randomization

CONTACTS AND LOCATIONS:
Overall Officials: Chen Chao, PhD,MD, Study Director — Chiledren's Hospital of Fudan University
Locations (3):
- China (3):
  - Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided